CLINICAL TRIAL: NCT04820036
Title: A Physiologic Analysis of Endoscopic Sleeve Gastroplasty (ESG): Effects of ESG on Non-Alcoholic Steatohepatitis (NASH) and Portal Pressure Gradient in Patients With Obesity and NASH With Advanced Fibrosis
Brief Title: A Physiologic Analysis of Endoscopic Sleeve Gastroplasty (ESG)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Pichamol Jirapinyo, MD, MPH, Associate Director of Bariatric Endoscopy, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020P003540
Record Dates: First submitted 2021-03-17; First posted 2021-03-29 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Non-alcoholic Steatohepatitis (NASH); Endoscopic Sleeve Gastroplasty; Non-alcoholic Fatty Liver Disease (NAFLD); Endoscopic Ultrasound; Liver Function; Obesity; Liver Fibroses
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Liver Cirrhosis | interventions — Liver Function Tests

STUDY DESIGN:
Intervention Model Description: Prospective pilot observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients with Obesity and NASH scheduled/recommended for P-ESG Procedure (Other): We will perform a 12-month prospective, single-center, pilot observational study on patients with obesity and NASH with advanced fibrosis who are undergoing P-ESG. A total of 15 patients will undergo EUS-LB with EUS-PPG measurement in a single session prior to and at 12 months following P-ESG
  Interventions: Diagnostic Test: Insulin Resistance; Behavioral: Quality of Life Assessment; Diagnostic Test: Liver Function Test; Diagnostic Test: Radiologic features of NASH; Diagnostic Test: Serologic features of NASH

INTERVENTIONS:
Diagnostic Test: Insulin Resistance — Insulin resistance: Fasting glucose and insulin will also be measured to calculate Homeostatic Model Assessment of Insulin Resistance (HOMA-IR), as a surrogate of IR
Behavioral: Quality of Life Assessment — Quality of life will be assessed using the Chronic Liver Disease Questionnaire.
Diagnostic Test: Liver Function Test — EUS-guided liver biopsy and portal pressure gradient measurement
Diagnostic Test: Radiologic features of NASH — Controlled attenuation parameter (CAP) and liver stiffness scores assessed by transient elastography (TE)
Diagnostic Test: Serologic features of NASH — Laboratory value assessment of alanine aminotransferase (ALT), liver chemistries, platelet counts, albumin and calculated NAFLD Fibrosis Score (NFS).

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is the most common chronic liver disease worldwide. Affecting approximately one-third of the United States (U.S.) population, the prevalence of NAFLD increases to 90% in patients with obesity. In 25% of patients, NAFLD progresses to a more severe form-non-alcoholic steatohepatitis (NASH)-which further increases the risks of cirrhosis and hepatocellular carcinoma. In 2017, the lifetime costs of caring for NASH patients in the U.S. were estimated at $222.6 billion, with the cost of caring for the advanced NASH (fibrosis stage ≥ 3) being $95.4 billion. It is projected that the number of NASH cases will increase by 63% from 2015 to 2030. Given the weight loss efficacy of Endoscopic Bariatric and Metabolic Therapies (EBMTs), it has been suggested that EBMTs may serve as a novel treatment category for NASH. Previously, the PI and Co-Is studied the effect of Intragastric balloons (IGB)-the oldest EBMT device-on NASH. EUS liver biopsy performed at the time of IGB removal revealed resolution of all NASH histologic features including fibrosis. A follow-up study by a different group showed similar findings. Furthermore, studies have showed the benefits of S-ESG and Aspiration Therapy (AT) on non-histologic features of NASH. Given the greater weight loss experienced after P-ESG compared to IGB (20% vs 10% TWL) and the more reproducible technique and shorter learning curve of the current P-ESG compared to S-ESG, we aim to assess the effect of P-ESG on NASH.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is the most common chronic liver disease worldwide. Affecting approximately one-third of the United States (U.S.) population, the prevalence of NAFLD increases to 90% in patients with obesity. In 25% of patients, NAFLD progresses to a more severe form-non-alcoholic steatohepatitis (NASH)-which further increases the risks of cirrhosis and hepatocellular carcinoma. In 2017, the lifetime costs of caring for NASH patients in the U.S. were estimated at $222.6 billion, with the cost of caring for the advanced NASH (fibrosis stage ≥ 3) being $95.4 billion. It is projected that the number of NASH cases will increase by 63% from 2015 to 2030.

Liver biopsy (LB) remains the gold standard for diagnosing NASH. Although the presence of fibrosis is not required for diagnosis, fibrosis stage is the strongest predictor of liver-related outcomes, with stages 3 and 4 being associated with a mortality relative risk of 6.7 and 11.1, respectively, compared to no fibrosis. Traditionally, LB has been performed via a percutaneous or transjugular approach. With advancements in endoscopic ultrasound (EUS) technologies, EUS-guided LB (EUS-LB) has emerged as an alternative means, with a 90%-100% diagnostic yield and 0-0.9% adverse event (AE) rate.

In patients with advanced fibrosis, the main determinant of decompensation and mortality is the presence of portal hypertension (PH), defined as hepatic venous portal gradient (HVPG) > 5 mmHg. In 2017, Dr. Guadalupe Garcia-Tsao (Co-I) further subcategorized compensated cirrhosis into those with no PH (HVPG ≤ 5 mmHg), mild PH (HVPG > 5 but < 10 mmHg) and clinically significant PH (HVPG ≥ 10 mmHg) given the differences in their pathophysiological mechanisms, prognosis and potentially therapeutic approach.

Traditionally, HVPG is obtained by subtracting the free hepatic venous pressure (FHVP) from the wedged hepatic venous pressure (WHVP), which is used as a surrogate of portal venous pressure (PVP). In 2016, Dr. Marvin Ryou (Co-I) reported the safety and technical feasibility of measuring true PVP and HVP and thus directly assess portal pressure gradient (PPG) in pigs using a digital pressure wire delivered through an EUS-based needle. Since then, the technology has progressed with the current device consisting of an EUS-based needle connected to a digital compact manometer. Studies in humans now report 92%-100% technical success without AEs (compared to 7-9% AE rate for traditional LB).

The mainstay of treatment for NASH remains weight loss achieved via lifestyle modification (LM). Previous studies show a correlation between weight loss and improvement in histologic features of NASH with approximately 10% total weight loss (TWL) required for fibrosis regression. Nevertheless, the average weight loss associated with LM is 3.8%, with less than 10% of patients able to achieve the 10% TWL threshold, leaving the majority of NASH patients undertreated.

Endoscopic bariatric and metabolic therapy (EBMT) is an emerging field for the treatment of obesity. To date, four EBMT devices/procedures are approved by the Food and Drug Administration (FDA) and available: intragastric balloon (IGB), endoscopic sleeve gastroplasty via suturing (S-ESG), endoscopic sleeve gastroplasty via plication (P-ESG), also known as POSE, and aspiration therapy (AT).

P-ESG involves the use of an endoscopic plication device to reduce gastric volume. While P-ESG has been available in the U.S. for almost a decade, in 2017, Dr. Christopher Thompson (Co-I) invented a new plication pattern. Specifically, instead of placing plications primarily in the fundus, a novel P-ESG procedure, also known as distal POSE, involves placing plications in the gastric body, sparing the fundus. In addition to assisting with the first new P-ESG case in 2017, the PI, along with Dr. Thompson, has continued to refine the techniques to optimize efficiency, efficacy and generalizability. With the current technique, P-ESG appears reproducible and associated with a shorter learning curve compared to S-ESG. Furthermore, our study estimated a mean of 15% TWL, with all patients achieving ≥ 10% TWL without AEs at 6 months and a mean of 20% TWL at 12 months (see Preliminary Data).

Given the weight loss efficacy of EBMTs, it has been suggested that EBMTs may serve as a novel treatment category for NASH. Previously, the PI and Co-Is studied the effect of IGB-the oldest EBMT device-on NASH. EUS-LB performed at the time of IGB removal revealed resolution of all NASH histologic features including fibrosis. A follow-up study by a different group showed similar findings. Furthermore, studies have showed the benefits of S-ESG and AT on non-histologic features of NASH. Given the greater weight loss experienced after P-ESG compared to IGB (20% vs 10% TWL) and the more reproducible technique and shorter learning curve of the current P-ESG compared to S-ESG, we aim to assess the effect of P-ESG on NASH.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18-65 years old
* Obesity (defined as BMI > 30 kg/m2)
* Biopsy-proven NASH (defined as the presence of steatosis and hepatic injury in the form of ballooning or lobular inflammation)19
* Advanced fibrosis (defined as bridging fibrosis (F3) or cirrhosis (F4) on LB).

Exclusion Criteria:

* Decompensated cirrhosis (defined as bleeding varices, ascites, encephalopathy and jaundice)
* gastric varices
* diabetes mellitus (defined as HbA1c ≥ 6.5%)
* active smoking
* being on an anticoagulant or anti-platelet medication
* active participation in any weight loss program, the use of a weight loss medication over the past 6 months and history of bariatric surgery or EBMT.
* Patients with esophageal varices are not excluded as long as they are on a non-selective beta-blocker for primary prophylaxis.
* Patient is pregnant, breast-feeding, or planning to become pregnant during the course of the study.
* Patient is unwilling or unable to sign and date the informed consent.
* Patient is unwilling or unable to comply with the follow-up study schedule.
* Patient for whom endoscopic procedures are contraindicated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2027-12-24 (Estimated)

PRIMARY OUTCOMES:
Change in Month 0 liver function at 12 months. | Month 0, Month 12
  EUS-guided liver biopsy with portal pressure gradient measurement

SECONDARY OUTCOMES:
Change in Month 0 radiologic features of NASH at 6 and 12 months. | Month 0, Month 6, Month 12
  Assessed using controlled attenuation parameter (CAP) and Liver Stiffness scores assessed by transient elastography (TE).
Change in Month 0 serologic features of NASH at 6 and 12 months. | Month 0, Month 6, Month 12
  Assessed by laboratory assessment of liver enzymes and calculating NAFLD Fibrosis Score (NFS) ((calculated using age, body mass index (BMI), liver chemistries, platelet counts and albumin)
Change in Month 0 Anthropometric factors at months 1,3,6,9,12. | Months 0, Month 1, Month 3, Month 6, Month 9, Month 12
  Assessment of weight, waist circumference, body composition measured at every follow-up visit
Change in Month 0 insulin resistance at 6 and 12 months. | Month 0, Month 6, Month 12
  Fasting glucose and insulin will also be measured to calculate Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Change in Month 0 Quality of Life at 12 months. | Month 0, Month 12
  This will be assessed using the "Chronic Liver Disease Questionnaire" (CLDQ-NASH). The instrument includes 36 items grouped into 6 domains: Abdominal Symptoms, Activity/Energy, Emotional Health, Fatigue, Systemic Symptoms, and Worry. In CLDQ-NASH, patients are asked about how frequently they experience certain problems impairing various aspects of their well-being; a 1-7 Likert scale is used for the responses (the score of 1 would correspond to a problem is experienced "All of the time", and the score of 7 to "None of the time"). The final scoring scheme suggests that the scores are calculated separately for each domain as an average of the domain's items. In all domains, greater scores reflect better health, and the average of the domain scores yields the total CLDQ-NASH score.

CONTACTS AND LOCATIONS:
Overall Officials: Pichamol Jirapinyo, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Formal contract for data sharing will need to be executed with the Institution prior to sharing with other researchers.